CLINICAL TRIAL: NCT03752138
Title: Phase I Study of TK216 in Patients With Relapsed and Refractory Leukemias
Brief Title: TK216 and Decitabine in Treating Patients With Relapsed and Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The supporting pharamceutical company elected not to pursue this study at this time.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0495; NCI-2018-02667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0495 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 Part 1 TK216: Days 1-7 (Experimental): Patients receive TK216 IV continuously on days 1-7 every 21 days.
  Interventions: Drug: Group 1: TK216
- Group 2 Part 1 TK216: Days 1-7 and 15-28 (Experimental): Patients receive TK216 IV on days 1-7 and 15-21 every 28 days.
  Interventions: Drug: Group 2: TK216
- Part 2 TK216 + Decitabine 10mg/m2 (Experimental): Patients receive recommended dose of TK216 from Part 1 plus Decitabine.
  Interventions: Drug: Part 2: Decitabine 10mg/m2; Drug: Part 2: TK216
- Part 2 TK216 + Decitabine 20 mg/m2 (Experimental): Patients receive recommended dose of TK216 from Part 1 plus Decitabine.
  Interventions: Drug: Part 2: Decitabine 20 mg/m2; Drug: Part 2: TK216
- Expansion Phase: TK216 + Decitabine (Experimental): All patients in the expansion cohort will receive the RP2D of TK216 and Decitabine.
  Interventions: Drug: Expansion Phase TK216; Drug: Expansion Phase Decitabine

INTERVENTIONS:
Drug: Group 1: TK216 — Starting Dose: 288 mg/m2 given by vein on Days 1-7 of a 21 day cycle.
  Arms: Group 1 Part 1 TK216: Days 1-7
Drug: Group 2: TK216 — Starting Dose: 144 mg/m2 given by vein on Days 1-7 and 15-21 of a 23 day cycle.
  Other Names: TK-216; TK216
  Arms: Group 2 Part 1 TK216: Days 1-7 and 15-28
Drug: Part 2: Decitabine 10mg/m2 — 10mg/m2 by vein on Days 1-10 of a 28 day cycle.
  Other Names: Dacogen
  Arms: Part 2 TK216 + Decitabine 10mg/m2
Drug: Part 2: Decitabine 20 mg/m2 — 20 mg/m2 by vein on Days 1-10 of a 28 dayi cycle.
  Other Names: Dacogen
  Arms: Part 2 TK216 + Decitabine 20 mg/m2
Drug: Expansion Phase TK216 — Expansion cohort will receive the RP2D of TK216
  Arms: Expansion Phase: TK216 + Decitabine
Drug: Expansion Phase Decitabine — Expansion cohort will receive the RP2D of Decitabine
  Other Names: Dacogen
  Arms: Expansion Phase: TK216 + Decitabine
Drug: Part 2: TK216 — Recommended dose from Part 1.
  Arms: Part 2 TK216 + Decitabine 10mg/m2; Part 2 TK216 + Decitabine 20 mg/m2

SUMMARY:
This phase I trial studies the side effects and best dose of TK216 and decitabine when given together in treating patients with acute myeloid leukemia that has come back or does not respond to treatment. Drugs used in chemotherapy, such as TK216 and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLT) of Ets-family transcription factor inhibitor TK216 (TK216) in patients with relapsed and refractory (R/R) acute myeloid leukemia (AML). (Phase I Dose Escalation) II. To determine the safety and tolerability of TK216 combined with decitabine in patients with relapsed and refractory AML. (Combination Cohort)

SECONDARY OBJECTIVES:

I. Safety profile of TK216 as characterized by adverse event (AE) type, severity, timing and relationship to study drug, as well as laboratory abnormalities in the first and subsequent treatment cycles. (Phase I Dose Escalation) II. To explore the efficacy (complete remission [CR], complete remission without platelet recovery [CRp], complete remission without blood count recovery [CRi], or partial remission [PR]), of TK216 as a single-agent in patients with R/R AML. (Phase I Dose Escalation) III. To assess overall survival (OS), and disease free survival (DFS) in patients with R/R AML treated with TK216. (Phase I Dose Escalation) IV. Duration of disease control defined as first date of disease control identified (either CR/CRp/CRi, PR or SD) until the date of progression. (Phase I Dose Escalation) V. To explore biomarkers of response and resistance in patients with R/R AML treated with TK216. (Phase I Dose Escalation) VI. Safety profile of TK216 in combination with decitabine as characterized by adverse event (AE) type, severity, timing and relationship to study drug, as well as laboratory abnormalities in the first and subsequent treatment cycles. (Combination Cohort) VII. To explore the efficacy (complete remission [CR], complete remission without platelet recovery [CRp], complete remission without blood count recovery [CRi], or partial remission [PR], of TK216 in combination with decitabine in patients with R/R AML. (Combination Cohort) VIII. To assess overall survival (OS), and progression free survival (PFS) in patients with R/R AML treated with TK216 + decitabine. (Combination Cohort) IX. Duration of disease control defined as first date of disease control identified (either CR/CRp/CRi, PR or SD) until the date of progression. (Combination Cohort) X. To explore biomarkers of response and resistance in patients with R/R AML treated with TK216 + decitabine. (Combination Cohort)

OUTLINE: This is a dose-escalation study.

Patients receive TK216 intravenously (IV) continuously on days 1-7 every 21 days, or continuously on days 1-7 and 15-21 every 28 days. Patients also receive decitabine IV over 60 minutes on days 1-10 every 28 days. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of histologically confirmed relapsed or refractory (R/R) acute myeloid leukemia for which no available standard therapies are indicated or anticipated to result in a durable response
* Patients must not have had leukemia therapy for 14 days prior to starting TK216. However, patients with rapidly proliferative disease may receive hydroxyurea as needed until 24 hours prior to starting therapy on this protocol and during the first cycle of study
* Bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 3 x upper limit of normal (ULN) -- or =< 5 x ULN if related to leukemic involvement
* Creatinine =< 1.5 x ULN
* Known cardiac ejection fraction of > or = 45% within the past 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* A negative urine pregnancy test is required within 1 week for all women of childbearing potential prior to enrolling on this trial
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol

Exclusion Criteria:

* Pregnant women are excluded from this study because the agent used in this study has the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided
* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient with documented hypersensitivity to any of the components of the therapy program
* Patients with active, uncontrolled central nervous system (CNS) leukemia will not be eligible
* Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use at least 1 form of barrier birth control (such as condom) prior to study entry and for the duration of study participation
* Patients with known history of serous retinopathy will not be eligible
* Prior treatment with TK216

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-31 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days
  Will be tabulated with frequency and percentage by grade, attribution to treatment, and by dose level/schedule.
Response rate | Up to 30 days
  Will be estimated alone with 95% confidence interval.
Overall survival | Up to 1 year
  Will be estimated using the Kaplan-Meier method.
Disease free survival | Up to 1 year
  Will be estimated using the Kaplan-Meier method.
Duration of disease control | Up to 1 year
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Kadia, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org